CLINICAL TRIAL: NCT00612456
Title: A Double-masked, Randomized, Parallel-group Study to Investigate the Pharmacodynamics, Safety, and Systemic Pharmacokinetics of Pazopanib Drops, Administered for 28 Days to Adult Subjects With Neovascular Age-related Macular Degeneration.
Brief Title: To Evaluate the Pharmacodynamics, Safety, and Pharmacokinetics of Pazopanib Drops in Adult Subjects With Neovascular AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD7108240
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2017-09-28 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-09

CONDITIONS: Macular Degeneration
Keywords: angiogenesis; pazopanib,; age-related macular degeneration (AMD),; vascular endothelial growth factor (VEGF),; choroidal neovascularization (CNV),
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Pazopanib eye drops formulation 5 mg/mL daily for 28 days
  Interventions: Drug: Pazopanib
- Arm 2 (Experimental): Pazopanib eye drop formulation 5mg/mL TID for 28 days
  Interventions: Drug: Pazopanib
- Arm 3 (Experimental): Pazopanib eye drop formulation 2mg/mL TID for 28 days
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib eye drops formulation

SUMMARY:
This is a 28 day study to evaluate the pharmacodynamic effect of pazopanib eye drops on the central retinal thickness of AMD patients

DETAILED DESCRIPTION:
Pazopanib has been formulated as an eye drop for the topical treatment of age-related macular degeneration (AMD). Safety, tolerability and pharmacokinetics have been evaluated in a first study conducted in healthy volunteers (MD7108238). In the present study, three dosing regimens of pazopanib eye drops, administered for 28 days, will be evaluated in subjects with occult or minimally classic subtypes of choroidal neovascularization due to AMD. This study is designed to measure pharmacological activity of topically administered pazopanib in target tissues (choroid and retina) of patients with AMD by weekly evaluation of central retinal thickness as measured by optical coherence tomography (OCT). Evaluation of efficacy will be performed on an exploratory basis by weekly measurement of visual acuity. The ocular and systemic safety and systemic pharmacokinetics of pazopanib treatment for 28 days will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age-related macular degeneration patients diagnosed with subfoveal choroidal neovascularization in the study eye, with all of the following characteristics required:

  * central subfield thickness > 300 microns on investigator-determined OCT (inclusive of subretinal fluid)
  * active subfoveal leakage as determined by investigator-determined fluorescein angiography
  * minimally classic or occult with no classic CNV lesion
  * lesion size no greater than 12 disc areas
  * CNV > 50% of lesion area
  * < 50% of lesion area with blood
  * = 25% of lesion area with fibrosis
* Best-corrected ETDRS visual acuity in the study eye between 80 to 24 letters inclusive (approximately 20/25 and 20/320 or 4/5 to 4/63) at screening
* Female subjects must be of non-childbearing potential.

Exclusion Criteria:

* Additional eye disease in the study eye that could compromise best corrected visual acuity (i.e. glaucoma with documented visual field loss, clinically significant diabetic retinopathy, ischemic optic neuropathy, or retinitis pigmentosa).
* CNV in the study eye due to other causes unrelated to age-related macular degeneration.
* The presence of retinal angiomatous proliferation (RAP) in the study eye, as determined by the investigator (confirmation by indocyanine green angiography is not required).
* Geographic atrophy involving the center of the fovea in the study eye.
* Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation of the fundus for photographs, fluorescein angiography and OCT.
* Vitreous, subretinal or retinal hemorrhage in the study eye that is unrelated to AMD.
* More than one prior photodynamic therapy (PDT) treatment in the study eye.
* PDT treatment in the study eye < 12 weeks prior to dosing.
* Previous treatment in the study eye with ranibizumab (Lucentis) or bevacizumab (Avastin) without resolution of exudation (intraretinal and subretinal fluid as documented by OCT).
* Use of any treatment, either approved or experimental, for AMD in the study eye within 60 days of first dose of investigational product.
* Intraocular surgery in the study eye within 3 months of dosing.
* Aphakia or total absence of the posterior capsule (Yttrium aluminum garnet (YAG) capsulotomy permitted) in the study eye.
* History of vitrectomy in the study eye.
* Use of topical ocular medications in the study eye within 7 days of first dose of investigational product or expected use of topical ocular medications during the treatment period, with the exception of artificial tears (refer to Section 9.1)
* Active treatment in the fellow eye, with the exception of preservative-free artificial tears.
* Current use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol).
* Use of systemic steroids (>10 mg prednisone or equivalent/day) within 14 days of first dose.
* An unwillingness to refrain from wearing contact lenses starting from the screening visit, through the follow-up visit
* Medical history or condition:

  * Uncontrolled Diabetes Mellitus, with hemoglobin A1c (HbA1c) > 10%.
  * Myocardial infarction or stroke within 12 months of screening.
  * Active bleeding disorder.
  * Major surgery within 1 month of screening.
  * Hepatic impairment.
* Uncontrolled hypertension

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-03-05 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2009-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (16):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Winter Haven, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Australia (3):
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Perth, Western Australia
- GSK Investigational Site, Leuven, Belgium
- Italy (5):
  - GSK Investigational Site, Trieste, Friuli Venezia Giulia
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 22 centers in the United States, Belgium, Italy and Australia between 18 February 2008 and 27 January 2009. A total of 70 participants with Age-related macular degeneration (AMD) were randomized to the study.
Groups:
- Pazopanib 5 mg/mL TID: Eligible participants received Pazopanib eye drops topically at a dose of 5 milligrams per milliliter (mg/mL) three time daily (TID) for 28 days. Participants were instructed to administer drops with a 6-hour interval between daily doses.
- Pazopanib 2 mg/mL TID: Eligible participants received Pazopanib eye drops topically at a dose of 2 mg/mL TID for 28 days. Participants were instructed to administer drops with a 6-hour interval between daily doses.
- Pazopanib 5 mg/mL Once Daily: Eligible participants received Pazopanib eye drops topically at a dose of 5 mg/mL once daily for 28 days. Participants were instructed to administer drops with a 6-hour interval between daily doses.
Period: Overall Study
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Started | 27 | 27 | 16
Completed | 25 | 25 | 16
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pazopanib 5 mg/mL TID: Eligible participants received Pazopanib eye drops topically at a dose of 5 mg/mL TID for 28 days. Participants were instructed to administer drops with a 6-hour interval between daily doses..
- Total: Total of all reporting groups
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily | Total
Number analyzed (Participants) | 27 | 27 | 16 | 70
Age, Customized [Count of Participants; unit: Participants]
  57 to 88 years | 27 | 27 | 16 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 9 | 43
  Male | 7 | 13 | 7 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 27 | 27 | 16 | 70
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Central Retinal/Lesion Thickness (CRLT) as Measured by the Carl Zeiss Meditec Stratus Optical Coherence Tomography (OCT) Scanner at Day 29
Description: CRLT was measured by the Carl Zeiss Meditec Stratus OCT scanner based on the manual measurement of the distance between the inner and outer retina, inclusive of subretinal fluid and any choroidal neovascularization (CNV) as measured in the central 1 millimeter (mm) area of the 7 mm Posterior Pole Scan. OCT scans/images were collected by trained and certified photographer and analyzed by investigator. Two datasets were used for analysis namely Last observation carried forward (LOCF) which included missing assessment for a participant who completed at least 7 days of pazopanib eye drop replaced by the last non-missing assessment post 7 days of pazopanib eye drop treatment. OC dataset included a missing assessment at any scheduled time was considered unevaluable and was not imputed. Baseline was defined as the assessments performed between Day -3 to -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization value at Day 29.
Time Frame: Baseline (Day -3 to -1) and Day 29
Population: Pharmacodynamics (PD) parameters population comprised of all participants in the Safety Population and had Choroidal Neovascularization (CNV) present as detected by Fluorescein Angiography (FA). LOCF and OC dataset were used for analysis. Only those participants with data available at the indicated time point were included for analysis.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 26 | 24 | 14
Microns
  CRLT as measued by OCT, LOCF data | 7.5 (110.34) | 10.0 (83.78) | 31.2 (85.72)
  CRLT as measued by OCT, OC data: number analyzed (Participants) | 26 | 21 | 11
  CRLT as measued by OCT, OC data | 7.5 (110.34) | 3.0 (85.16) | 9.1 (69.12)
Statistical Analysis 1: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means using the LOCF dataset; p = 0.6241, ANCOVA — If the estimates of change from baseline in CRLT were negative, then the one-sided p-values were the two-sided t-test of each treatment arm from this analysis divided by 2. If the estimates of change from baseline in CRLT were positive, then the one; Mean Difference (Final Values) = 5.83, 95% CI 2-sided [-31.05 to 42.71], Standard Error of Mean 18.332
Statistical Analysis 2: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means using the LOCF dataset; p = 0.7315, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.87, 95% CI 2-sided [-26.52 to 50.26], Standard Error of Mean 19.081
Statistical Analysis 3: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means using the OC dataset; p = 0.6212, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.76, 95% CI 2-sided [-31.65 to 43.18], Standard Error of Mean 18.566
Statistical Analysis 4: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means using the OC dataset; p = 0.5987, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.20, 95% CI 2-sided [-36.44 to 46.84], Standard Error of Mean 20.662
Statistical Analysis 5: Comparison: Pazopanib 5 mg/mL TID; LOCF Data excluding potential one outlier participant. Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.4820, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -0.82, 95% CI 2-sided [-37.28 to 35.64], Standard Error of Mean 18.114
Statistical Analysis 6: Comparison: Pazopanib 2 mg/mL TID; LOCF Data excluding potential one outlier participant. Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.8562, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 19.90, 95% CI 2-sided [-17.33 to 57.13], Standard Error of Mean 18.496
Statistical Analysis 7: Comparison: Pazopanib 5 mg/mL TID; OC Data excluding potential one outlier participant. Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.4880, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-37.46 to 36.35], Standard Error of Mean 18.300
Statistical Analysis 8: Comparison: Pazopanib 2 mg/mL TID; OC Data excluding potential one outlier participant. Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.7556, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 13.97, 95% CI 2-sided [-26.38 to 54.32], Standard Error of Mean 20.008

2. Secondary Outcome: Number of Participants With Complete Ophthalmic Examination Values of Potential Clinical Concern
Description: A complete eye examination was performed to include the following: Examination of eyelids and lashes (including meibomian glands), Pupil, motility and confrontation visual field examination, Slit lamp evaluation of anterior ocular structures (including conjunctiva, tear film, cornea with fluorescein staining, anterior chamber, iris, lens, and anterior vitreous), intraocular pressure (IOP) measurement and Dilated Fundus Examination (Indirect ophthalmoscopy and slit lamp biomicroscopy). Data has been presented in a consolidated format for the total number of participants with values of potential clinical concern for complete ophthalmic examinations until Day 43.
Time Frame: Upto follow-up (Day 43)
Population: Safety population comprised of all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Pazopanib 5 mg/mL TID: Eligible participants received Pazopanib eye drops topically at a dose of 5 mg/mL TID for 28 days. Participants were instructed to administer drops approximately with a 6-hour interval between daily doses.
- Pazopanib 2 mg/mL TID: Eligible participants received Pazopanib eye drops topically at a dose of 2 mg/mL TID for 28 days. Participants were instructed to administer drops approximately with a 6-hour interval between daily doses.
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 27 | 27 | 16
Participants | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Vital Sign Data for Systolic Blood Pressure and Diastolic Blood Pressure and Heart Rate of Potential Clinical Concern
Description: Vital sign assessments included systolic blood pressure, diastolic blood pressure and heart rate. The potential clinical concern range for systolic blood pressure was <85 and > 160 millimeters of mercury, diastolic blood pressure <45 and > 100 millimeters of mercury, heart rate <40 and >110 beats per minute. Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important findings at any visit were reported.
Time Frame: Up to follow up (Day 46)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 27 | 27 | 16
Participants
  Systolic blood pressure | 1 | 4 | 1
  Diastolic blood pressure | 0 | 1 | 0
  Heart rate | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings
Description: Single 12-lead ECGs were to be obtained at each Day 15 and follow-up Day 43 using an ECG machine that automatically calculated the heart rate and measures PR, QRS, QT, and QTc intervals. ECG findings were defined as abnormal-not clinically significant (A-NCS) and abnormal-clinically significant (A-CS). Data has been presented for the number of participants with A-NCS and A-CS findings.
Time Frame: Day 15 and follow-up (Day 43)
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 27 | 27 | 16
Participants
  Day 15, A-NCS: number analyzed (Participants) | 27 | 26 | 16
  Day 15, A-NCS | 11 | 11 | 6
  Day 15, A-CS: number analyzed (Participants) | 27 | 26 | 16
  Day 15, A-CS | 1 | 0 | 0
  Follow-up (Day 43), A-NCS: number analyzed (Participants) | 26 | 27 | 16
  Follow-up (Day 43), A-NCS | 7 | 10 | 8
  Follow-up (Day 43), A-CS: number analyzed (Participants) | 26 | 27 | 16
  Follow-up (Day 43), A-CS | 2 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinical Chemistry and Hematology Data of Potential Clinical Concern
Description: Clinical chemistry parameters assessed included blood urea nitrogen, potassium, calcium, albumin, creatinine, chloride, sodium, total protein, glucose, total carbon dioxide, aspartate amino transferase, alanine amino transferase, direct bilirubin, total bilirubin, alkaline phosphatase and hematology parameters assessed included platelet count, white blood cell count, red blood cell count, reticulocyte count, hemoglobin, mean corpuscle volume, mean corpuscle hemoglobin, mean corpuscle hemoglobin concentration, total neutrophils, lymphocytes, monocytes, eosinophils, basophils. Data has been presented for the number of participants with values high and low of potential clinical concern for clinical chemistry and hematology.
Time Frame: Up to follow-up Day 43
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 27 | 27 | 16
Participants
  Glucose high | 4 | 1 | 1
  Glucose low | 2 | 0 | 0
  Calcium low | 1 | 0 | 0
  Potassium high | 1 | 1 | 0
  Total bilirubin high | 1 | 0 | 0
  Alkaline phosphatase high | 1 | 0 | 0
  Lymphocytes low | 1 | 1 | 1
  Total neutrophils low | 0 | 0 | 1

6. Secondary Outcome: Number of Participants With Abnormal Urinalysis Data by Dipstick Analysis
Description: Urinalysis included analysis for urine occult blood, urine glucose, urine ketones and urine proteins via dipstick analysis. Data has been presented for number of participants with abnormal urinalysis results. Only categories with values have been presented.
Time Frame: Day 29 and follow-up (Day 43)
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 27 | 27 | 16
Participants
  Urine Occult Blood at Day 29 1 hour, 1+: number analyzed (Participants) | 27 | 25 | 16
  Urine Occult Blood at Day 29 1 hour, 1+ | 1 | 1 | 2
  Urine Occult Blood at Day 29 1 hour, 2+: number analyzed (Participants) | 27 | 25 | 16
  Urine Occult Blood at Day 29 1 hour, 2+ | 0 | 1 | 0
  Urine Occult Blood at Follow-up, 1+: number analyzed (Participants) | 26 | 26 | 16
  Urine Occult Blood at Follow-up, 1+ | 1 | 0 | 0
  Urine Glucose at Day 29 1 hour, 1+ OR 1/4: number analyzed (Participants) | 27 | 25 | 16
  Urine Glucose at Day 29 1 hour, 1+ OR 1/4 | 0 | 1 | 1
  Urine Glucose at Follow-up, 3+ OR 1 gram/deciliter: number analyzed (Participants) | 26 | 26 | 16
  Urine Glucose at Follow-up, 3+ OR 1 gram/deciliter | 0 | 0 | 1
  Urine Protein at Day 29 1 hour, 1+: number analyzed (Participants) | 27 | 25 | 16
  Urine Protein at Day 29 1 hour, 1+ | 2 | 2 | 1
  Urine Protein at Day 29 1 hour, 2+: number analyzed (Participants) | 27 | 25 | 16
  Urine Protein at Day 29 1 hour, 2+ | 0 | 1 | 0
  Urine Protein at Follow-up, 1+: number analyzed (Participants) | 26 | 26 | 16
  Urine Protein at Follow-up, 1+ | 0 | 2 | 0
  Urine Protein at Follow-up, 3+: number analyzed (Participants) | 26 | 26 | 16
  Urine Protein at Follow-up, 3+ | 0 | 1 | 0

7. Secondary Outcome: Number of Participants With Ocular Adverse Events, Non-ocular Adverse Events, Serious Ocular Adverse Events and Serious Non-ocular Adverse Events
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury. Data has been presented for number of participants with ocular and non-ocular adverse events and serious adverse event
Time Frame: Up to follow-up (Day 43)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 27 | 27 | 16
Participants
  Non-Ocular Adverse Events | 10 | 5 | 2
  Ocular Adverse Events, Fellow eye | 2 | 0 | 1
  Ocular Adverse Events, Study eye | 9 | 2 | 3
  Non-Ocular Serious Adverse Events | 0 | 1 | 0

8. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) [Number of Letter Read on Standardized Early Treatment of Diabetic Retinopathy Study (ETDRS) Charts at Day 29
Description: BCVA was measured in the study eye using the ETDRS grading charts consists of at least 24 to 78 letters placed at a test distance of 4 meters. There were 7 cut off points in visual acuity on ETDRS grading chart: 15 to 29, 10 to 14, 5 to 9, -4 to 4, -5 to -9, -10 to -14 and -15 to -29 letters. Grade 15 to 29 indicates no impairment in vision and grade -15 to -29 indicates worst impairment in vision. Analyses were done for two sub-efficacy-populations. One sub-efficacy population included all participants in the efficacy population with a YES for retinal angiomatous proliferation (RAP)/retinal choroidal anastomosis (RCA) NONE field from Digital angiography reading center (DARC) FA form in study eye. The other included all participants in the efficacy population with a YES for eligible field from DARC FA form in study eye. Baseline was defined as the assessments performed between Day -3 to -1. Change from Baseline calculated as subtracting the Baseline value from the value at Day 29.
Time Frame: Baseline (Day -3 to -1) and Day 29
Population: Efficacy population comprised of all participants in the Safety Population who completed at least 7 days of pazopanib eye drop treatment and provided VA measurements and had CNV present as detected by FA. Only those participants available at the specified time points were included for analysis.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 26 | 24 | 14
Scores on scale
  BCVA at Day 29: number analyzed (Participants) | 26 | 22 | 11
  BCVA at Day 29 | 4.3 (5.95) | 0.8 (8.38) | 0.0 (2.05)
  YES for RAP/RCA NONE field from DARC FA at Day 29: number analyzed (Participants) | 25 | 21 | 10
  YES for RAP/RCA NONE field from DARC FA at Day 29 | 4.8 (5.67) | 1.7 (7.43) | -0.1 (2.13)
  YES for eligible field from DARC FA form at Day 29: number analyzed (Participants) | 19 | 18 | 7
  YES for eligible field from DARC FA form at Day 29 | 3.5 (5.26) | 0.8 (7.39) | 0.3 (1.38)
Statistical Analysis 1: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means based on efficacy population; p = 0.0015, ANCOVA; Mean Difference (Final Values) = 4.32, 95% CI 2-sided [1.74 to 6.91], Standard Error of Mean 1.290
Statistical Analysis 2: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means based on efficacy population; p = 0.5921, ANCOVA; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-2.05 to 3.57], Standard Error of Mean 1.403
Statistical Analysis 3: Comparison: Pazopanib 5 mg/mL Once Daily; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means based on efficacy population; p = 0.9646, ANCOVA; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-3.89 to 4.07], Standard Error of Mean 1.988
Statistical Analysis 4: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means based on participants with a 'YES' for RCA NONE field from DARC FA form in study eye at screening; p = 0.0003, ANCOVA; Mean Difference (Final Values) = 4.75, 95% CI 2-sided [2.32 to 7.19]
Statistical Analysis 5: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — [test comment as in outcome 8, analysis 4]; p = 0.2208, ANCOVA; Mean Difference (Final Values) = 1.64, 95% CI 2-sided [-1.02 to 4.30], Standard Error of Mean 1.326
Statistical Analysis 6: Comparison: Pazopanib 5 mg/mL Once Daily; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — [test comment as in outcome 8, analysis 4]; p = 0.9847, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-3.90 to 3.83], Standard Error of Mean 1.927
Statistical Analysis 7: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — Statistics has been presented for least square means based on participants with a 'YES' for eligible field from DARC FA form in study eye at screening; p = 0.0142, ANCOVA; Mean Difference (Final Values) = 3.53, 95% CI 2-sided [0.75 to 6.31], Standard Error of Mean 1.376
Statistical Analysis 8: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — [test comment as in outcome 8, analysis 7]; p = 0.5547, ANCOVA; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-2.02 to 3.71], Standard Error of Mean 1.419
Statistical Analysis 9: Comparison: Pazopanib 5 mg/mL Once Daily; Comparison between Baseline value and Day 29 value; Test type: Superiority or Other — [test comment as in outcome 8, analysis 7]; p = 0.9114, ANCOVA; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-4.37 to 4.88], Standard Error of Mean 2.287

9. Secondary Outcome: Number of Participants With Change in Retinal Morphology (Cystoid Spaces, Subretinal Fluid and Retinal Pigment Epithelial Detachment) as Determined by OCT
Description: OCT was used for the determination of retinal morphology changes in the study eye which included assessments of cystoids spaces (cyst like spaces in the inner layers of the retina), subretinal fluid (an exudate between the retina and choroid from various sources including the vitreous cavity, subarachnoid space, or abnormal vessels) and pigment epithelial detachment (retinal pigment epithelium separates from the underlying Bruch's membrane due to the presence of blood, serous exudate, drusen, or a neovascular membrane). Data has been presented for number of participants with retinal morphology changes in the study eye at Day 29.
Time Frame: Day 29
Population: PD Parameter Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 26 | 21 | 11
Participants
  Cystoid spaces at Day 29 | 9 | 10 | 5
  Pigment epithelial detachment at Day 29 | 1 | 2 | 1
  Subretinal fluid at Day 29 | 2 | 4 | 2

10. Secondary Outcome: Number of Participants With Change in Characteristics (Fibrosis, Atrophy, Blood) as Measured by Fundus Photography (FP)
Description: Fundus photography involves capturing of images of the center of the very back inner wall of the eye - the retina, optic nerve, macula and main retinal blood vessels. The parameters assessment were heme subretinal hemorrhage (absence or presence at the location), heme intraretinal hemorrhage (absence or presence at the location), subretinal fluid (absence or presence at location), fibrosis (absence or presence at location), atrophy (absence or presence of atrophic changes) and pigment ((absence or presence at location). A protocol set of fundus photographs were obtained at Day 29. Images were read by the investigator for eligibility determination, and by a central reading center for determination of PD effect. Data has been presented for number of participants with changes in eye characteristics in the study eye at Day 29.
Time Frame: Day 29
Population: PD Parameter Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 26 | 22 | 11
Participants
  Heme subretinal hemorrhage at Day 29 | 14 | 14 | 7
  Heme intraretinal hemorrhage at Day 29 | 7 | 1 | 1
  Subretinal fluid at Day 29 | 26 | 22 | 11
  Fibrosis at Day 29 | 2 | 2 | 1
  Atrophy at Day 29 | 6 | 6 | 5
  Pigment at Day 29 | 23 | 20 | 11

11. Secondary Outcome: Change From Baseline in Neovascular Size, Total Lesion Size, Fluorescein Angiography (FA) Leakage Area of Measurement, FA Blood Area of Measurement as Measured by FA at Day 29
Description: FA uses FP to capture images of injected dye circulating throughout the retinal blood vessels to assess leaking, swelling or circulation problems caused by various eye diseases like diabetic retinopathy and wet macular degeneration. The parameters assessed were CNV size, Classic CNV size, FA blood area of measurement, FA leakage area of measurement and total lesion size. A protocol fluorescein angiogram was to be obtained at Day 29. Images were evaluated by investigator for eligibility determination, and by a central reading center for determination of PD effect. Data has been presented for change from baseline in change in eye characteristics in the study eye at Day 29. Baseline was defined as the assessments performed between Day -3 to -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization value at Day 29.
Time Frame: Baseline (Day -3 to -1) and Day 29
Population: PD Parameter Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
Number analyzed (Participants) | 26 | 24 | 14
millimeters
  CNV size at Day 29: number analyzed (Participants) | 25 | 22 | 10
  CNV size at Day 29 | 0.6 (1.67) | 0.44 (2.04) | 0.7 (1.96)
  Classic CNV size at Day 29: number analyzed (Participants) | 6 | 4 | 3
  Classic CNV size at Day 29 | 0.2 (0.90) | 1.5 (1.62) | 0.7 (0.81)
  FA blood area of measurement at Day 29: number analyzed (Participants) | 10 | 7 | 5
  FA blood area of measurement at Day 29 | -0.2 (0.75) | 1.0 (1.87) | 0.4 (0.82)
  FA leakage area of measurement at Day 29: number analyzed (Participants) | 25 | 22 | 10
  FA leakage area of measurement at Day 29 | 0.8 (1.77) | 0.8 (2.06) | 0.6 (1.88)
  Total lesion size: number analyzed (Participants) | 25 | 22 | 11
  Total lesion size | 0.5 (1.57) | 1.2 (2.37) | 0.7 (1.86)
Statistical Analysis 1: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value for FA Leakage Area of measurement; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.0534, ANCOVA; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-0.01 to 1.53], Standard Error of Mean 0.383
Statistical Analysis 2: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value for FA Leakage Area of measurement; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.0508, ANCOVA; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.00 to 1.64], Standard Error of Mean 0.409
Statistical Analysis 3: Comparison: Pazopanib 5 mg/mL Once Daily; Comparison between Baseline value and Day 29 value for FA Leakage Area of measurement; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.3141, ANCOVA; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.60 to 1.83]
Statistical Analysis 4: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value for FA Blood Area of measurement; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.6018, ANCOVA; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.04 to 0.62], Standard Error of Mean 0.395
Statistical Analysis 5: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value for FA Blood Area of measurement; Test type: Superiority or Other; p = 0.0509, ANCOVA — Statistics has been presented for least square means; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [-0.00 to 2.00], Standard Error of Mean 0.476
Statistical Analysis 6: Comparison: Pazopanib 5 mg/mL Once Daily; Comparison between Baseline value and Day 29 value for FA Blood Area of measurement; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.3976, ANCOVA; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.70 to 1.68], Standard Error of Mean 0.566
Statistical Analysis 7: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value for Total Lesion size; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.2410, ANCOVA; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-0.32 to 1.23], Standard Error of Mean 0.385
Statistical Analysis 8: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value for Total Lesion size; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.0032, ANCOVA; Mean Difference (Final Values) = 1.27, 95% CI 2-sided [0.44 to 2.09], Standard Error of Mean 0.412
Statistical Analysis 9: Comparison: Pazopanib 5 mg/mL Once Daily; Comparison between Baseline value and Day 29 value for Total Lesion size; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.3185, ANCOVA; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-0.58 to 1.75], Standard Error of Mean 0.581
Statistical Analysis 10: Comparison: Pazopanib 5 mg/mL TID; Comparison between Baseline value and Day 29 value for CNV Size; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.1074, ANCOVA; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.14 to 1.37], Standard Error of Mean 0.377
Statistical Analysis 11: Comparison: Pazopanib 2 mg/mL TID; Comparison between Baseline value and Day 29 value for CNV Size; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.0403, ANCOVA; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [0.04 to 1.65], Standard Error of Mean 0.402
Statistical Analysis 12: Comparison: Pazopanib 5 mg/mL Once Daily; Comparison between Baseline value and Day 29 value for CNV Size; Test type: Superiority or Other — Statistics has been presented for least square means; p = 0.2490, ANCOVA; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-0.50 to 1.88], Standard Error of Mean 0.594

12. Secondary Outcome: Plasma Pharmacokinetic Parameter Maximum Observed Concentration (Cmax)
Description: Blood samples for analysis of plasma pazopanib concentrations were collected over 6 hours after an ocular dose of pazopanib on Day 15 or Day 22. PK analyses of plasma pazopanib concentration-time data were conducted using non-compartmental Model 200 (for extravascular administration) of WinNonlin Professional Edition version 5.2. Data has been presented for pharmacokinetic parameter Cmax at Day 15 and Day 22.
Time Frame: Day 15 and Day 22
Population: The pharmacokinetic population included all participants in the Safety Population who received at least one dose of active treatment and a PK sample was obtained and analyzed. Only those participants available at the specified time points were used for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID
Number analyzed (Participants) | 24 | 24
nanograms per milliliter
  Day 15: number analyzed (Participants) | 24 | 23
  Day 15 | 56.104 (85.38) | 21.142 (75.53)
  Day 22: number analyzed (Participants) | 0 | 1
  Day 22 |  | 17.680 (NA) — Geometric coefficient variation could not be calculated as only a single participant was analyzed.

13. Secondary Outcome: Plasma Pharmacokinetic Parameter Time of Occurrence of Cmax (Tmax)
Description: Blood samples for analysis of plasma pazopanib concentrations were collected over 6 hours after an ocular dose of pazopanib on Day 15 or Day 22. PK analyses of plasma pazopanib concentration-time data were conducted using non-compartmental Model 200 (for extravascular administration) of WinNonlin Professional Edition version 5.2. Data has been presented for pharmacokinetic parameter tmax at Day 15 and Day 22.
Time Frame: Day 15 and Day 22
Population: Pharmacokinetic population. Only those participants available at the specified time points were used for analysis.
Measure: Median (Full Range); unit: hour
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID
Number analyzed (Participants) | 24 | 24
hour
  Day 15: number analyzed (Participants) | 24 | 23
  Day 15 | 3.000 [0.00 to 6.00] | 2.970 [0.00 to 6.42]
  Day 29: number analyzed (Participants) | 0 | 1
  Day 29 |  | 3.000 [3.00 to 3.00]

14. Secondary Outcome: Plasma Pharmacokinetic Parameter Area Under Concentration Time-curve From Time Zero to 6 Hours (AUC [0-6)]
Description: Blood samples for analysis of plasma pazopanib concentrations were collected over 6 hours after an ocular dose of pazopanib on Day 15 or Day 22. PK analyses of plasma pazopanib concentration-time data were conducted using non-compartmental Model 200 (for extravascular administration) of WinNonlin Professional Edition version 5.2. Data has been presented for pharmacokinetic parameter AUC (0-6) at Day 15 and Day 22.
Time Frame: Day 15 and Day 22
Population: Pharmacokinetic population. Only those participants available at the specified time points were used for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per hour per milliliter
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID
Number analyzed (Participants) | 24 | 24
nanograms per hour per milliliter
  Day 15: number analyzed (Participants) | 22 | 21
  Day 15 | 312.17998 (87.87) | 124.57714 (77.00)
  Day 22: number analyzed (Participants) | 0 | 1
  Day 22 |  | 96.13500 (NA) — Geometric coefficient variation could not be calculated as only a single participant was analyzed.

ADVERSE EVENTS:
Time Frame: Up to follow-up (Day 43)
Description: Safety population was used for analysis.
Arm/Group | Pazopanib 5 mg/mL TID | Pazopanib 2 mg/mL TID | Pazopanib 5 mg/mL Once Daily
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/27 | 0/16
Other Adverse Events (participants affected / at risk) | 7/27 | 1/27 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 5 mg/mL TID (N=27) | Pazopanib 2 mg/mL TID (N=27) | Pazopanib 5 mg/mL Once Daily (N=16)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 5 mg/mL TID (N=27) | Pazopanib 2 mg/mL TID (N=27) | Pazopanib 5 mg/mL Once Daily (N=16)
Retinal disorder (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 1
Myodesopsia (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.